CLINICAL TRIAL: NCT02743884
Title: Prospective, Interventional Study Evaluating Heat Transfer With the Esophageal Cooling Device
Brief Title: Evaluating Heat Transfer With the Esophageal Cooling Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, d sessler, Chair Department of Outcomes Research, The Cleveland Clinic
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 16-124
Record Dates: First submitted 2016-04-14; First posted 2016-04-19 (Estimated); Last update posted 2017-04-13 (Actual); Status verified 2017-04

CONDITIONS: Non-cardiac Surgery

STUDY DESIGN:
Intervention Model Description: Cross-over.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Esophageal Cooling Device (Experimental): Esophageal cooling
  Interventions: Device: Esophageal Cooling
- Esophageal Warming (Experimental): Esophageal warming
  Interventions: Device: Esophageal Warming

INTERVENTIONS:
Device: Esophageal Warming — 30 minutes of warming from circulating water at about 42 degrees C through an esophageal heat exchanger.
  Arms: Esophageal Warming
Device: Esophageal Cooling — 30 minutes of cooling from circulating water at about 7 degrees C through an esophageal heat exchanger.
  Arms: Esophageal Cooling Device

SUMMARY:
An esophageal heat exchange tube will be inserted in anesthetized surgical patients. Each patient will have 30 minutes of cooling (circulating fluid at 7 degrees C) and 30 minutes of warming (42 degrees C) with 15-minute recovery break in between. The primary outcome will be heat transfer, determined from inflow and outflow temperatures and fluid flow rate for cooling and warming modes.

DETAILED DESCRIPTION:
The ECD is made with medical-grade silicone and has 3 ports; 2 coolant ports and a central port. The coolant ports of the ECD are connected to external heat exchanger while a third, central lumen simultaneously allows gastric decompression and drainage. The ECD can be inserted like a standard gastric tube.

The aim of this prospective, interventional study is to quantify heat transfer during warming and cooling using the Esophageal Cooling Device in anesthetized patients having non-cardiac surgery.

An esophageal heat exchange tube will be inserted in anesthetized surgical patients. Each will have 30 minutes of cooling (circulating fluid at 7 degrees C) and 30 minutes of warming (42 degrees C) with 15 -minute break in between; the order of the cooling and warming will be randomized. The primary outcome will be heat transfer, determined from inflow and outflow fluid temperatures and fluid flow rate assessed for both cooling and warming modes.

ELIGIBILITY:
Inclusion Criteria:

* Elective non-cardiac surgery;
* Age 18-80 years;
* Surgery expected to last >2 hours;
* General anesthesia with endotracheal Intubation;
* Volatile anesthesia;
* BMI < 38 kg/m2;
* ASA physical status 1-3.

Exclusion Criteria:

* Weight < 45 kg;
* Unstable blood pressure;
* Known esophageal deformity or evidence of esophageal trauma or esophageal disease that in the opinion of the attending anesthesiologist precludes safe use of ECD.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Mean heat transfer at cooling, kcal/h | 15-60 minutes after intubation during elective non-cardiac surgery
  Heat transfer is calculated as difference between inflow and outflow temperatures, multiplied by flow and the specific heat of water
Mean heat transfer at warming, kcal/h | 15-60 minutes after intubation during elective non-cardiac surgery
  Heat transfer is calculated as difference between inflow and outflow temperatures, multiplied by flow and the specific heat of water

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Sessler, M.D., Study Chair — Dept Chairman
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No